CLINICAL TRIAL: NCT02118688
Title: Efficacy and Safety of Risperidone and Trazodone Monotherapy and Combination Therapy in Critically Ill Patients With Delirium: A Four-arm Prospective, Randomized, Double-blind, Placebo-controlled Pilot Study
Brief Title: Efficacy and Safety of Risperidone and Trazodone Monotherapy and Combination Therapy in Critically Ill Patients With Delirium
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, Mindee S. Hite, Critical Care Clinical Pharmacy Specialist, Rochester General Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICUDelirium
Record Dates: First submitted 2014-04-09; First posted 2014-04-21 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Delirium; Agitation
MeSH Terms: conditions — Delirium; Psychomotor Agitation | interventions — Risperidone; Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Drug: Placebo
  * Placebo suspension administered PO/NG/FT q12h to mimic risperidone
  * Placebo suspension administered PO/NG/FT q8h to mimic trazodone
  Interventions: Drug: Placebo
- Risperidone alone (Active Comparator): Drug: Risperidone
  * Initiate risperidone at 1 mg PO/NG/FT q12h
  * Risperidone dose can be titrated upwards every 24 hours by increments of 0.5 mg per dose
  * Maximum risperidone daily dose of 6 mg per day (3 mg every 12 hours)
  Interventions: Drug: Risperidone; Drug: Placebo
- Trazodone alone (Active Comparator): Drug: Trazodone
  * Initiate trazodone dosing at 50 mg PO/NG/FT q8h
  * Trazodone dose can be titrated upwards every 24 hours by 25 mg per dose
  * Maximum trazodone daily dose 600 mg per day (200 mg every 8 hours)
  Interventions: Drug: Trazodone; Drug: Placebo
- Risperidone and Trazodone combination (Active Comparator): Drug: Risperidone
  * Initiate risperidone at 1 mg PO/NG/FT q12h
  * Risperidone dose can be titrated upwards every 24 hours by increments of 0.5 mg per dose
  * Maximum risperidone daily dose of 6 mg per day (3 mg every 12 hours)
  Drug: Trazodone
  * Initiate risperidone at 1 mg PO/NG/FT q12h
  * Risperidone dose can be titrated upwards every 24 hours by increments of 0.5 mg per dose
  * Maximum risperidone daily dose of 6 mg per day (3 mg every 12 hours)
  Interventions: Drug: Risperidone; Drug: Trazodone

INTERVENTIONS:
Drug: Risperidone
  Arms: Risperidone alone; Risperidone and Trazodone combination
Drug: Trazodone
  Arms: Risperidone and Trazodone combination; Trazodone alone
Drug: Placebo
  Arms: Placebo; Risperidone alone; Trazodone alone

SUMMARY:
The purpose of this randomized clinical trial is to determine whether risperidone alone, trazodone alone, or a combination of risperidone and trazodone is superior for the treatment of ICU acquired delirium. The hypothesis is that combination therapy is superior to either agent alone in treating ICU acquired delirium and sustaining delirium free time.

DETAILED DESCRIPTION:
Delirium is defined as a disturbance of consciousness characterized by an acute onset of impaired cognitive function. Although delirium is thought to be common in the Intensive Care Unit (ICU) there are few studies that have evaluated its incidences, risks and outcomes. It has been associated with increased morbidity, and mortality and increased cost to the healthcare system. In addition to the uncertainty of the incidence of ICU delirium, there is a lack of information about the effects that certain pharmacological treatments have on delirious patients.

The rationale for this study is to evaluate the efficacy and safety of risperidone alone, trazodone alone, and risperidone plus trazodone for the treatment of delirium in critically ill patients when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old who are admitted for more than 24 hours in the MICU or SICU
* Patients diagnosed with delirium by primary team (screened positive for delirium using the CAM-ICU or with clinical manifestations of delirium)
* Patients have an order for as-needed haloperidol or have received a one-time dose of haloperidol within 24 hours of randomization
* Patients must be tolerating enteral feeding (greater than 20 mL/hour for more than 12 hours)

Exclusion Criteria:

* Patients who are unlikely to survive 24 hours after admission to the ICU
* Patients who are admitted with a primary neurological condition or injury (i.e. stroke, active seizures, prolonged coma, overdose)
* Patients who can not actively participate in delirium assessment
* Patients actively withdrawing from alcohol or narcotics
* Patients who were treated with any antipsychotic or trazodone within 30 days prior to ICU admission
* Patients with a marked baseline prolongation of the QTc interval (repeated demonstration of QTc interval greater 500 milliseconds (msec))
* Patients with a history of Torsades de Pointes
* Patients with current treatment with an agent having either the potential to affect or increase the risk of QTc prolongation (e.g. erythromycin, any class Ia, Ic, or III antiarrhythmics)
* Patients being treated with a neuromuscular blocker
* Patients in whom haloperidol, risperidone, or trazodone is contraindicated
* Pregnant patients or patients who are breast-feeding
* Patients with a modified Blessed dementia rating scale score ≥4 or an Informant Questionnaire of Cognitive Dysfunction in the Elderly Score ≥4
* Patients in which informed consent can not be obtained from the legally authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The number of days patients are without delirium during the study period (delirium-free days) | Every 24 hours (up to 14 days)
  The number of days patients are without delirium during the study period (delirium-free days)

SECONDARY OUTCOMES:
Daily prevalence of delirium as indicated by a positive Confusion Assessment Method in the ICU (CAM-ICU) | Every 24 hours (up to 14 days)
Resolution of delirium as indicated by a negative Confusion Assessment Method in the ICU (CAM-ICU) for more than 24 hours | Every 24 hours (up to 14 days)
The number of patients who require rescue medications, the type of rescue medications utilized, and the amount of rescue medications per day | Every 24 hours (up to 14 days)
The number of patients who receive sedative agents, amount of midazolam equivalents per day, and the number of days in which patients receive a sedative agent | Every 24 hours (up to 14 days)
The number of patients who receive pain medications, amount of fentanyl equivalents per day, and the number of days in which patients receive a pain medication | Every 24 hours (up to 24 hours)
The number of hours spent agitated (RASS score between +4 and +2) as a percent of the time that the study drug was administered | Every 24 hours (up to 14 days)
The number of hours spent excessively sedated or in a coma state (RASS score between -4 to -5) as a percent of the time that the study drug was administered | Every 24 hours (up to 14 days)
The duration of mechanical ventilation from initial intubation to extubation as long as the patient remained extubated for more than 48 hours. | Time (hours) from initial intubation to extubation (as long as patient not reintubated within 48 hours)
The number of days that the patients were alive and breathing without assistance during the study period (ventilator-free days) | Time (days) from extubation to patient discharge (as long as patient not reintubated within 48 hours)
The number of episodes and number of patients who experience clinically significant QTc prolongation (≥ 500 msec or an increase of more than 60 msec from baseline) | QTc interval evaluated q12h during period of study drug administration (up to 14 days)
The number of episodes and number of patients who experience clinically significant extrapyramidal effects (as evidenced by a positive Simpson-Angus Scale Score) | Extrapyramidal effects evaluated by bedside nurse q12h during period of study drug administration (up to 14 days). Investigator will confirm RN suspicion of extrapyramidal effects using Simpson-Angus Score.
All-cause mortality and 28-day mortality | At 14 and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mindee S Hite, Pharm.D., Principal Investigator — Rochester General Hospital
Locations (1):
- Rochester General Hospital, Rochester, New York, United States